CLINICAL TRIAL: NCT06462859
Title: Effect of Sensory Integration on Motor Function, Balance, and Trunk Control in Diplegic Cerebral Palsy
Brief Title: Effect of Sensory Integration in Diplegic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Halic University (Other)
Responsible Party: Principal Investigator, Ayşen Canan Pakeloğlu, MSc Student, Halic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HalicU-FTR-ACP-01
Record Dates: First submitted 2024-06-11; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Diplegic Cerebral Palsy
Keywords: Cerebral Palsy; Diplegia Type; Treatment; Balance
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Two groups with a neurodevelopmental treatment control group
Who Masked: Participant, Outcomes Assessor
Masking Description: Information regarding the allocation of each group was not provided and outcome assessment was performed by an investigator blinded to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group (Experimental): The experimental group received sensory integration therapy in addition to the NDT program.Both groups participated in NDT sessions for 45 minutes, three times a week, over a span of 8 weeks.
  Interventions: Other: Sensory Integration Therapy Group; Other: Neurodevelopmental Treatment Group
- Control Group (Other): The NDT program was customized for each child, incorporating a unique blend of static and dynamic balance exercises, coordination exercises, mobility exercises, and strength training exercises.Both groups participated in NDT sessions for 45 minutes, three times a week, over a span of 8 weeks.
  Interventions: Other: Neurodevelopmental Treatment Group

INTERVENTIONS:
Other: Sensory Integration Therapy Group — The experimental group received sensory integration therapy in addition to the NDT program. The NDT program is customized for each child, featuring a unique blend of static and dynamic balance exercises, coordination exercises, mobility exercises, and strength training exercises. Participants attended 45-minute NDT and sensory integration sessions three times a week for 8 weeks. Sensory integration therapy, visual perception activities (block design, shape recognition in pictures, puzzles, matching geometric shapes and letters, numbers and classification exercises), body awareness activities (showing body parts, drawing life-size drawings, turning left and right, recognizing body parts by touching ), tactile perception exercises (feeling and touching various textures and shapes) and visual-motor coordination training (eye tracking exercises, activities with moving objects and panel activities).
  Arms: The experimental group
Other: Neurodevelopmental Treatment Group — The NDT program is customized for each child, featuring a mix of static and dynamic balance exercises, coordination exercises, mobility exercises, and strength training exercises. He attended 45-minute NDT sessions three times a week for 8 weeks. There is no treatment or medication other than NDT.

SUMMARY:
The purpose of this study is to compare the effects of sensory integration therapy (SIT) applied in addition to neurodevelopmental treatment (NDT) on Motor Function, Balance, and Trunk Control in diplegia cerebral palsy

DETAILED DESCRIPTION:
Cerebral palsy is the most frequent motor disability affecting children. The condition is characterized by problems with postural control and balance, which are due to the central nervous system being compromised by a brain lesion.

In sensory processing, the steps include receiving, organizing, and interpreting sensory information, followed by generating an appropriate response. Children develop motor skills through sensory experiences. Sensory integration therapy leads to enhanced body awareness, motor planning abilities, and coordination between both sides of the body.

Literature studies have demonstrated the effectiveness of sensory integration therapy in improving motor functions in children with diplegia type CP. However, there is a notable lack of research on how sensory integration therapy, in addition to neurodevelopmental treatment (NDT), affects balance and trunk control in these children. This study aims to bridge this gap by evaluating the impact of sensory integration therapy on gross motor function, balance, and trunk control in children with diplegia type CP when used as an adjunct to NDT.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between the ages of 4 and 17.
* Participants must be classified as Level II, III, or IV according to the Gross Motor Function Classification System (GMFCS).

Exclusion Criteria:

* Participants who had previously received sensory integration therapy, - Undergone Botulinum Toxin-A injections, or surgical interventions in the past year.
* Participants who were using pharmacological agents affecting muscle tone.
* Participants with an uncontrolled history of epilepsy.
* Participants who were unable to attend the study regularly.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Measure-88 (GMFM-88) | 8 weeks
  The evaluation is organized into sections based on different motor skills: Section A covers lying and rolling, Section B includes sitting, Section C focuses on crawling and kneeling, Section D assesses standing, and Section E includes walking, running, and jumping. Altogether, there are 88 items: Section A (17 items), Section B (20 items), Section C (14 items), Section D (13 items), and Section E (24 items). The minimum clinically important difference (MCID) ranges from 0.8 to 1.6 for a medium effect size and 1.3 to 2.6 for a larger effect size.

SECONDARY OUTCOMES:
Pediatric Balance Scale (PBS) | 8 weeks
  The PBS includes 14 items designed to assess daily life activities and functional skills. Each section is scored from 0 to 4, with a maximum total score of 56. A higher score indicates better functional balance performance.
Trunk Control Measurement Scale (TCMS) | 8 weeks
  This assessment includes 15 items where children follow commands to perform movements within specific subsections, with their performance scored accordingly. The total score ranges from 0 to 58, with higher scores denoting better trunk control. The items gauge gross motor functions by assessing the child's performance. Each section is rated on a 4-point Likert scale, and percentages are calculated for each section. The final score is obtained by summing these percentages and dividing by 5.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşen Canan Pakeloğlu, MSc, Principal Investigator — Halic University; Seda Saka, Asst. Prof., Principal Investigator — Halic University
Locations (1):
- Ziya Special Education and Rehabilitation Center, Istanbul, Kagıthane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No